CLINICAL TRIAL: NCT06012565
Title: KAND567 Versus Placebo in Subjects Hospitalized With COVID-19. A Phase II, Randomized, 2-Arm Parallel-Group, Double-blind Study to Evaluate Efficacy, Safety, Tolerability, and Pharmacokinetics
Brief Title: KAND567 Versus Placebo in Subjects Hospitalized With COVID-19
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Novakand Pharma AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KAN0006; 2020-002322-85 (EudraCT Number)
Record Dates: First submitted 2023-08-24; First posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — microcrystalline cellulose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Statistician and Safety Review Committee are not blinded. Sponsor is blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KAND567 (Experimental)
  Interventions: Drug: KAND567
- Placebo (Placebo Comparator)
  Interventions: Drug: Microcrystalline cellulose

INTERVENTIONS:
Drug: KAND567 — 2 x 125 mg capsules for oral administration. KAND567 (250 mg) was to be given every 12 hours for one week (7 days).
  Arms: KAND567
Drug: Microcrystalline cellulose — Capsules for oral administration, consisting of microcrystalline cellulose oral solid formulation in capsules. Placebo was to be given every 12 hours for one week (7 days).
  Arms: Placebo

SUMMARY:
The study is a phase II, randomized, 2-arm parallel-group, double-blind study to explore the efficacy, safety, tolerability and pharmacokinetics of KAND567 versus placebo in COVID-19 subjects in need of oxygen treatment.

The target was to include forty (40) subjects with diagnosed COVID-19 for participation in the study. If at screening all criteria for study participation were fulfilled and informed consent signed, the subject was enrolled and randomized into one of the two arms. After randomization, the subjects were to receive KAND567 or placebo treatment for 7 days.

After the treatment period the subjects returned to ordinary clinical follow-up, but a study follow-up visit was to be planned for Day 21 and 90.

ELIGIBILITY:
Inclusion Criteria:

* Written Informed Consent obtained and documented according to national/local regulations prior to any study-specific procedure.
* Males and females aged ≥18-85 years at the time of signing the informed consent form.
* Patients with symptoms and signs of SARS-CoV-2 infection according to the World Health Organization (WHO) case definition. Symptoms must include shortness of breath, with an onset which occurred ≤ 10 days before admission, and the COVID-19 diagnosis must be confirmed by laboratory testing (PCR-positive). In addition, moderately impaired oxygenation as demonstrated by oxygen saturation ≤ 93% but ≥ 87% on room air, or requiring 1-5 L/min of oxygen to obtain an oxygen saturation of ≥ 92%, and at least one of the following laboratory values:

(A) Ferritin: > 300 ng/mL for men and > 150 ng/mL for women. (B) C-reactive protein (CRP): ≥ 10 mg/L. (C) D-dimer elevated above the age-adjusted lower limit: (i) ≤ 50 years; < 0.5 mg/L FEU (Fibrinogen Equivalent Units). (ii) > 50 years; age-related, calculated as follows: 0.5 mg/L FEU + 0.01 mg/L FEU for every year over 50 (i.e., one who is 70 years old has thus a reference limit of < 0.7 mg/L FEU; one who is 90 years old has a reference limit of < 0.9 mg/L FEU).

* Able to swallow capsules
* Male subject must be willing to use condoms with spermicide, and if he has a fertile partner, she must use contraceptive methods with a failure rate of < 1% to prevent pregnancy. Male subjects must also refrain from donating sperm from the first dose until three months after dosing with investigational product (IP). Female subjects must be post-menopausal or use contraceptive methods with a failure rate of < 1% to prevent pregnancy.
* Willingness and ability to comply with study procedures, visit schedules, study restrictions and requirements.

Exclusion Criteria:

* Patient not committed to aggressive management. For example, the subject, the subject's family or primary physician are unwilling to accept that the subject is placed on mechanical ventilation; or in the case of an advanced directive to withhold life support, with the exception of cardiopulmonary resuscitation.
* A suspected, active bacterial, fungal, viral, or other infection (besides COVID 19).
* Alanine aminotransferase (ALAT) or aspartate aminotransferase (ASAT) > 2 times the upper limit of normal (ULN) detected at screening (per local lab) or suspected liver disease.
* Uncontrolled or untreated symptomatic arrhythmias, myocardial infarction within the last 6 weeks, or decompensated congestive heart failure.
* Any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant (e.g., compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments.
* Clinically verified pulmonary embolism
* Chronic use of oral corticosteroids for treatment of inflammatory disease
* Use of strong CYP3A4 inhibitors (e.g., azoleantifungals, macrolide antibiotics, protease inhibitors) or inducers (e.g., rifabutin and rifampicin) and drugs sensitive to CYP3A4 inhibition (e.g., benzodiazepines, certain statins [lovastatin and simvastatin], certain P2Y12 inhibitors [ticagrelor and clopidogrel]).
* Participation in another pharmaceutical clinical study.
* Subject who has received any investigational drug within the last 3 months before administration of the investigational medicinal product (IMP).
* Severe COVID-19 at randomization: requiring non-invasive or invasive mechanical ventilation or Intensive Care Unit (ICU) admission for any other cause than respiratory support.
* Patients judged not to be suitable for non-invasive monitoring of oxygen saturation because of impaired peripheral circulation or for other reasons.
* Active malignancy with or without treatment, except local basal cell carcinoma.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2020-10-11 (Actual); Primary Completion 2021-08-07 (Actual); Study Completion 2021-08-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of KAND567, as measured by the occurrence of adverse events (AEs) and serious adverse events (SAEs). | From the first IMP administration (Day 1) until the last follow-up visit (Day 90).

CONTACTS AND LOCATIONS:
Overall Officials: Mantas Okas, MD, PhD, Principal Investigator — Capio St. Görans Hospital
Locations (4):
- Denmark (2):
  - Hvidovre Hospital, Hvidovre
  - Odense University Hospital, Odense
- Sweden (2):
  - Capio St. Görans Hospital, Stockholm
  - Västmanlands Hospital, Västerås

IPD SHARING:
Plan to Share IPD: No